CLINICAL TRIAL: NCT00138281
Title: Influenza Immunity: Protective Mechanisms Against a Pandemic Respiratory Virus
Brief Title: Influenza Immunity Against Pandemic Respiratory Virus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-183
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-03

CONDITIONS: Influenza
Keywords: influenza, vaccine, respiratory virus, Fluzone, FluMist
MeSH Terms: conditions — Influenza, Human | interventions — FluMist; Influenza Vaccines

INTERVENTIONS:
Biological: FluMist
Biological: Fluzone

SUMMARY:
Sixty adults, ages 18-49, will be randomly assigned to receive either FluMist or Fluzone. Some of the subjects will have participated in previous studies for these 2 vaccines. The study will last 4 months with subject participation being 28 days. The purpose of this study is to measure immune response to the vaccinations.

DETAILED DESCRIPTION:
This is a Phase 4, single-center, study of the immune responses of adults to one of two licensed influenza vaccines (either inactivated vaccine given IM or live, attenuated vaccine given intranasally). The study will enroll up to 60 adults, ages 18-49, some of whom were immunized in the Years 1 and 2 studies. This study began Year 1 of this grant with a protocol testing the two vaccine products in their age-approved populations. FluMist is approved for use in healthy children and adolescents, 5-17 years of age, and healthy adults 18-49 years of age. Fluzone is approved for all age groups starting at 6 months of age. To match for age and to study the youngest children possible, the age cohorts of 5-9 and 18-49 years were chosen for initial Year 1 study. In 2003, 70 adults and 16 children were enrolled, randomized 1:1 to receive either FluMist or Fluzone and immunized. In 2004, 44 of the original 70 adults were re-immunized with the same preparation they received in 2003. In addition, studies were conducted in twenty-eight 6mos to 5yo children who all received Fluzone and in thirty-nine 5-9 yo children who were randomized 1:1 to receive either FluMist or Fluzone. For 2005, we propose to study in this protocol, adults from last year who agree to a third immunization plus as many new adults to add up to a total of 60. Blood samples will also be taken at Days 0, 7-9 and 28 to be analyzed for CD4 and CD8 T-cell, B-cell, NK-cell and homing receptor responses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult, aged 18-49 years who have or have not participated in the Year 1 protocol.
2. Willing to sign informed consent.
3. Availability for follow-up for the planned duration of the study at least 4 weeks after immunization.
4. Acceptable medical history by screening evaluation and brief clinical assessment.
5. Negative urine or serum pregnancy test for women of childbearing potential.
6. If the subject is female and of childbearing potential, she must use an acceptable contraception and not become pregnant for the duration of the study. (Acceptable contraception includes implants, injectables, combined oral contraceptives, effective intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner).

Exclusion Criteria:

1. History of immunodeficiency.
2. Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; diabetes mellitus; moderate to severe kidney impairment.
3. History of Guillain-Barré syndrome.
4. Malignancy, other than squamous cell or basal cell skin cancer.
5. Autoimmune disease.
6. History of asthma or reactive airways disease.
7. Chronic cardiovascular and pulmonary disorder.
8. Chronic metabolic diseases (including diabetes), renal dysfunction or hemoglobinopathies requiring regular medical follow-up or hospitalization during the preceding year.
9. Use of immunosuppressive medication. Corticosteroid nasal sprays are permissible.
10. Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol.
11. Inactivated vaccine 14 days prior to vaccination.
12. Live, attenuated vaccines within 60 days of study.
13. Use of investigational agents within 30 days prior to study.
14. Receipt of blood products or immunoglobulin in the past 6 months.
15. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment.
16. Acute febrile illness on the day of vaccination.
17. Pregnant or lactating women.
18. Known allergies to any component of the vaccine, including thimerosal.
19. History of allergy to eggs or egg products.
20. Any condition that, in the opinion of the investigator, might interfere with study objectives.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Primary Completion 2005-11 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States